CLINICAL TRIAL: NCT01210521
Title: Use of Vitamin D3 for the Treatment of Steroid Resistant Asthmatic Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor terminated study due to inability to enroll subjects.
Sponsor: Florida Atlantic University (Other)
Responsible Party: Principal Investigator, Patricia Keating, Research Assistant Professor, Florida Atlantic University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: WIRB1116133
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Asthma
Keywords: Asthmatic Patients; Vitamin D; Steroid Resistant Asthmatic Patients; cholecalciferol
MeSH Terms: conditions — Asthma | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prior to intervention with Vitamin D (No Intervention): Patients will be analyzed for clinical, serological and immunological parameters before starting the interventional drug, Vitamin D.
- Vitamin D Intervention (Active Comparator): Patients will be analyzed for clinical, serological and immunological parameters after one month taking Vitamin D.
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — Vitamin D, (2000IU) will be administered orally, once a day, for one month.
  Arms: Vitamin D Intervention

SUMMARY:
The purpose of this study is to determine the effects of vitamin D3 on severe asthmatic patients. Vitamin D3 may alter the response of these patients to conventional steroid therapy, making them more responsive to the latter form of treatment. Patients will be treated daily with an oral dose (2,000 IU) of vitamin D3 for one month and their clinical and serological parameters, and immune function, will be evaluated. Results from pre- and post-vitaminD3 treatment will be compared.

DETAILED DESCRIPTION:
Asthma is one of the most common chronic diseases in childhood and one of the leading causes of morbidity in children. Its incidence has been growing, especially in the Western, highly industrialized nations. Glucocorticoids are used for the treatment of many inflammatory and autoimmune diseases, among them asthma, because they can switch off genes that code for pro- inflammatory cytokines and chemokines. Unfortunately, there is a substantial group of severe asthma patients that are steroid resistant. In addition, they suffer from the long term side effects of systemic steroid use.

Vitamin D3 plays an important role in the maintenance of several organ systems and its deficiency causes multiple and complex dysfunctions for the organism. Vitamin D3 has been originally described to regulate calcemia by absorbing calcium in the intestine and by increasing re-absorption of calcium in the kidneys. Recent studies have shown the important effects of Vitamin D3 on many other systems, especially as a modulator of the immune system, and its deficiency has been linked to several autoimmune and inflammatory diseases such as multiple sclerosis, inflammatory bowel disease, lupus erythematosus, rheumatoid arthritis and asthma.

Vitamin D inhibits the dysregulated antibody synthesis that is seen in asthmatics. It inhibits the proliferation of immune cells that produce inflammatory substances, and conversely, vitamin D enhances the function and proliferation of regulatory cells, through the induction of IL-10 producing T regulatory cells, and a very effective group of T regulatory cells characterized as CD4+ CD25+ FoxP3+ . Dendritic cell (DC) function is also modulated by Vitamin D. 1,25(OH)2vitaminD3 appears to generate tolerogenic dendritic cells (DC) in vivo, as demonstrated in models of transplantation and autoimmune diseases. Immature/tolerogenic DCs induce development of T regulatory cells by several mechanisms, including production of IL-10 or TGF-beta. Vitamin D3 increases the glucocorticoid receptor expression in asthmatic patients' T cells. In an interesting study on an asthma mouse model, treatment with Vitamin D combined with immunotherapy resulted in increased production of the inhibitory cytokine IL-10 in lung tissue and increased levels of TGF-beta in serum.

Overall these studies and others, support the hypothesis that Vitamin D induces regulatory T cells that are crucial for the control of autoimmune diseases such as asthma.

In spite of this attractive conceptual link between the benefits of vitamin D and immune regulation in SR asthma, no study has presented clinical data, i.e., pulmonary functions, quality of life score, reduction in steroid dose and other medications, and indices of better asthma control. There is also a dearth of ex-vivo data in order to confirm or refute in-vitro results. There is very little data that characterizes the effects of vitamin D supplementation on immune cells, cytokines, and asthma mediators.

ELIGIBILITY:
Inclusion Criteria: Diagnosis of severe steroid resistant asthmatic as defined by the American Thoracic Society workshop 2000. Patients must have been diagnosed for at least one year prior to the study. Patients must exhibit one or more major criteria and two minor criteria from the following list to be included in the study:

Definition of Severe Asthma by American Thoracic Society Consensus (2000). Major Characteristics

In order to achieve control to a level of mild-moderate persistent asthma:

1. Treatment with continuous or near continuous (>50% of year) oral corticosteroids
2. Requirement for treatment with high-dose inhaled corticosteroids:

Drug Dose (µg/d) Dose (puffs/d)

1. Beclomethasone dipropionate. > 1,260. > 40 puffs (42 µg /inhalation).

   > 20 puffs (84 µg/inhalation)
2. Budesonide > 1,200 > 6 puffs
3. Flunisolide > 2,000 > 8 puffs
4. Fluticasone propionate > 880 > 8 puffs(110µg), >4puffs(220 µg)
5. Triamcinolone acetonide > 2,000 > 20 puffs

Minor Characteristics

1. Requirement for daily treatment with a controller medication in addition to inhaled corticosteroids, e.g., long-acting β-agonist, theophylline, or leukotriene antagonist
2. Asthma symptoms requiring short-acting β-agonist use on a daily or near daily basis
3. Persistent airway obstruction (FEV1,80% predicted; diurnal PEF variability >20%)
4. One or more urgent care visits for asthma per year
5. Three or more oral steroid "bursts" per year
6. Prompt deterioration with<25% reduction in oral or inhaled corticosteroid dose
7. Near fatal asthma event in the past Additional minor characteristics include : normal diffusing capacity and methacholine PC20 be less than 8mg.

Exclusion Criteria: Patients diagnosed with the following conditions will be excluded:

Vitamin D resistant rickets, chronic renal failure, hypercalcemia (secondary to hyperparathyroidism or malignancy), Chronic Obstructive Pulmonary Disease, severe malabsorption syndrome, sarcoidosis, patients taking cardiac glycosides for cardiac arrythmias.

Pregnant or nursing women, and smoking patients will be excluded.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Pulmonary Function Test | Six months
  A pulmonary function test or spirometry, measures lung function by determining the volume and flow of air that can be inhaled or exhaled. FEV1is determined.

SECONDARY OUTCOMES:
Concentration of Interleukin 10(IL-10),in serum. | One year
  The concentration of IL-10,in serum will be determined by ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: James X Hartmann, PhD, Principal Investigator — Florida Atlantic University

IPD SHARING:
Plan to Share IPD: No
Study withdrwan

REFERENCES:
- [Background] Litonjua AA. Childhood asthma may be a consequence of vitamin D deficiency. Curr Opin Allergy Clin Immunol. 2009 Jun;9(3):202-7. doi: 10.1097/ACI.0b013e32832b36cd. PMID 19365260
- [Background] Xystrakis E, Kusumakar S, Boswell S, Peek E, Urry Z, Richards DF, Adikibi T, Pridgeon C, Dallman M, Loke TK, Robinson DS, Barrat FJ, O'Garra A, Lavender P, Lee TH, Corrigan C, Hawrylowicz CM. Reversing the defective induction of IL-10-secreting regulatory T cells in glucocorticoid-resistant asthma patients. J Clin Invest. 2006 Jan;116(1):146-55. doi: 10.1172/JCI21759. Epub 2005 Dec 8. PMID 16341266
- [Background] Taher YA, van Esch BC, Hofman GA, Henricks PA, van Oosterhout AJ. 1alpha,25-dihydroxyvitamin D3 potentiates the beneficial effects of allergen immunotherapy in a mouse model of allergic asthma: role for IL-10 and TGF-beta. J Immunol. 2008 Apr 15;180(8):5211-21. doi: 10.4049/jimmunol.180.8.5211. PMID 18390702
- [Background] Peterlik M, Cross HS. Vitamin D and calcium insufficiency-related chronic diseases: molecular and cellular pathophysiology. Eur J Clin Nutr. 2009 Dec;63(12):1377-86. doi: 10.1038/ejcn.2009.105. Epub 2009 Sep 2. PMID 19724293
- [Background] Larche M. Regulatory T cells in allergy and asthma. Chest. 2007 Sep;132(3):1007-14. doi: 10.1378/chest.06-2434. PMID 17873195